CLINICAL TRIAL: NCT04056468
Title: Phase 1 Pharmacokinetics and Safety Study of Oral Mobocertinib in Subjects With Moderate or Severe Hepatic Impairment and Normal Hepatic Function
Brief Title: A Study to Evaluate Pharmacokinetics (PK) and Safety of Oral Mobocertinib in Participants With Moderate or Severe Hepatic Impairment (HI) and Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TAK-788-1008; U1111-1236-7377 (Registry Identifier: WHO)
Record Dates: First submitted 2019-08-13; First posted 2019-08-14 (Actual); Results first posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-01

CONDITIONS: Hepatic Impairment; Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — mobocertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Moderate HI (Child-Pugh B): Mobocertinib 40 mg (Experimental): Mobocertinib 40 milligram (mg), capsule, orally, a single dose on Day 1.
  Interventions: Drug: Mobocertinib
- Severe HI (Child-Pugh C): Mobocertinib 40 mg (Experimental): Mobocertinib 40 mg, capsule, orally, a single dose on Day 1.
  Interventions: Drug: Mobocertinib
- Normal Hepatic Function: Mobocertinib 40 mg (Experimental): Mobocertinib 40 mg, capsule, orally, a single dose on Day 1.
  Interventions: Drug: Mobocertinib

INTERVENTIONS:
Drug: Mobocertinib — Mobocertinib capsule.
  Other Names: AP32788; TAK-788

SUMMARY:
The purpose of this study is to characterize the single-dose plasma PK of mobocertinib and its active metabolites (AP32960 and AP32914) in participants with moderate and/or severe HI compared to matched-healthy participants with normal hepatic function.

DETAILED DESCRIPTION:
29-Apr-2020 Enrollment of new participants into this study was paused due to the COVID-19 situation. The duration of this pause was dependent on the leveling and control of the COVID-19 pandemic.

The drug being tested in this study is called mobocertinib. The study will assess the PK of single dose mobocertinib and its active metabolites (AP32960 and AP32914) in participants with moderate and/or severe HI compared to matched-healthy participants with normal hepatic function.

The study will enroll approximately 24 participants. Participants will be assigned to 1 of the following 3 treatment groups in a staggered manner based on their degree of hepatic impairment which will be determined based on Child-Pugh Score as follow:

* Moderate HI (Child-Pugh B): Mobocertinib 40 mg
* Severe HI (Child-Pugh C): Mobocertinib 40 mg
* Normal Hepatic Function: Mobocertinib 40 mg

Healthy participants with normal hepatic function will be recruited to match both moderate and severe HI by age (mean plus or minus [+-] 10 years), gender (+-2 participants per gender), and body mass index (BMI, mean +-10 percent [%]).

All participants will be asked to take single dose of mobocertinib on Day 1. The dose level for severe HI may be modified based on the previous results of approximately 3 moderate HI and healthy participants who completed up to Day 10 study procedures.

This multi-center trial will be conducted in the United States. The overall time to participate in this study is approximately 51 days. Participants will be contacted by telephone 30 days after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Healthy Participants

1. Continuous non-smoker or moderate smoker (less than or equal to (<=) 10 cigarettes/day or the equivalent) before screening. Participant must agree to consume no more than 5 cigarettes or equivalent/day from the 7 days prior to mobocertinib dosing and throughout the period of PK sample collection.
2. Body mass index (BMI) greater than or equal to (>=) 18.0 and <=39.0 kilogram per square meter (kg/m^2), at screening. Participants will be matched to hepatic impaired participants by BMI (mean plus minus [+-] 10%) at screening. At least 50% of the participants will be required to be of BMI >=18.0 and <=35.0 kg/m^2, at screening.
3. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or electrocardiograms (ECGs), as deemed by the Investigator or designee. Has liver function tests including alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), and total bilirubin within the upper limit of normal at screening and at check-in.
4. Creatinine clearance (estimated glomerular filtration rate [eGFR]) >=60 milliliter per minute per 1.73 square meter (mL/min/1.73 m^2) at screening.

Inclusion Criteria for Moderate or Severe HI Participants

1. Continuous non-smoker or moderate smoker (<=10 cigarettes/day or the equivalent) before screening. Participant must agree to consume no more than 5 cigarettes or equivalent/day from the 7 days prior to mobocertinib dosing and throughout the period of pharmacokinetic(s) (PK) sample collection.
2. BMI >=18.0 and <=39.0 kg/m^2, at screening. At least 50% of the participants will be required to be of BMI >=18.0 and <=35.0 kg/m^2, at screening.
3. Aside from HI, be sufficiently healthy for study participation based upon medical history, physical examination, vital signs, ECGs, and screening clinical laboratory profiles, as deemed by the Investigator or designee.
4. Creatinine clearance (eGFR) >=60 mL/min/1.73 m^2 at screening.
5. Chronic HI for at least 3 months before screening, and the HI must be stable, that is, no significant changes in hepatic function in the 30 days preceding screening (or since the last visit if within 6 months before screening) and treatment with stable doses of medication. Has a score on the Child-Pugh Class at screening as follows:

   * Moderate HI arm, Child-Pugh Class B: >=7 and <=9.
   * Severe HI arm, Child-Pugh Class C: >=10 and <=15.

Exclusion Criteria:

1. Positive results for COVID-19 at screening or check in.
2. Seated blood pressure is less than 90/40 millimeters of Mercury (mmHg) or greater than 150/95 mmHg at screening.
3. Seated heart rate is lower than 40 beats per minute (bpm) or higher than 99 bpm at screening.
4. Healthy participants: QTcF interval is >=450 msec in males or >=470 msec in females; Moderate or Severe HI participants: QTcF interval is greater than (>) 500 msec OR has ECG findings deemed abnormal with clinical significance by the Investigator or designee at screening.
5. Unable to refrain from or anticipates the use of any medication or substance (including prescription or over-the-counter, vitamin supplements, natural or herbal supplements) for the prohibited time period.
6. Been on a diet incompatible with the on-study diet, in the opinion of the Investigator or designee, within the 30 days prior to dosing and throughout the study.
7. Donation of blood or had significant blood loss within 56 days prior to dosing.
8. Plasma donation within 7 days prior to dosing.
9. Healthy participants: Positive result at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV); Moderate or Severe HI participants: Positive result at screening for HIV, HBsAg positive participants are allowed to enroll if hepatitis B virus (HBV) deoxyribonucleic acid (DNA) is below 1000 copies/milliliter (mL) in the plasma. Participants who are positive for hepatitis C virus antibodies (HCVAb) can be enrolled but must not have detectable HCV ribonucleic acid (RNA) in the plasma.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2022-02-05 (Actual); Study Completion 2022-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami, Hialeah, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in the United States from 09 October 2020 to 26 February 2022.
Pre-assignment Details: Participants with a diagnosis of moderate or severe hepatic impairment (HI) were enrolled to receive mobocertinib and were compared to a matched-normal hepatic function arm.
Period: Overall Study
Arm/Group | Moderate HI (Child-Pugh B): Mobocertinib 40 mg | Severe HI (Child-Pugh C): Mobocertinib 40 mg | Normal Hepatic Function: Mobocertinib 40 mg
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety set included all participants who received the study drug.
Groups:
- Moderate HI (Child-Pugh B): Mobocertinib 40 mg; Severe HI (Child-Pugh C): Mobocertinib 40 mg; Normal Hepatic Function: Mobocertinib 40 mg: Mobocertinib 40 mg, capsule, orally, a single dose on Day 1.
- Total: Total of all reporting groups
Arm/Group | Moderate HI (Child-Pugh B): Mobocertinib 40 mg | Severe HI (Child-Pugh C): Mobocertinib 40 mg | Normal Hepatic Function: Mobocertinib 40 mg | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (3.76) | 56.1 (8.64) | 59.4 (6.09) | 58.9 (6.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 7
  Male | 6 | 6 | 5 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 7 | 18
  Not Hispanic or Latino | 3 | 2 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 7 | 8 | 7 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 8 | 8 | 24
Weight [Mean (Standard Deviation); unit: kg] | 87.06 (24.847) | 81.46 (14.803) | 85.88 (16.824) | 84.80 (18.622)
Height [Mean (Standard Deviation); unit: cm] | 170.9 (11.72) | 169.4 (9.71) | 167.4 (8.98) | 169.2 (9.86)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI=weight/(height[m^2])
  kg/m^2 | 29.279 (4.7428) | 28.378 (4.5553) | 30.456 (4.0801) | 29.371 (4.3571)

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Mobocertinib and Its Active Metabolites (AP32960 and AP32914)
Time Frame: Day 1 pre-dose and at multiple time points (up to 216 hours) post-dose
Population: Pharmacokinetic (PK) set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile (e.g., exposure to treatment, availability of measurements and absence of major protocol violations).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Moderate HI (Child-Pugh B): Mobocertinib 40 mg | Severe HI (Child-Pugh C): Mobocertinib 40 mg | Normal Hepatic Function: Mobocertinib 40 mg
Number analyzed (Participants) | 8 | 8 | 8
nanograms per milliliter (ng/mL)
  Mobocertinib | 9.67 (58.2) | 11.3 (31.7) | 10.5 (37.6)
  AP32960 | 3.88 (28.8) | 2.82 (27.9) | 4.80 (23.6)
  AP32914 | 0.752 (38.6) | 0.722 (32.5) | 1.15 (31.7)

2. Primary Outcome: Cmax,u: Maximum Observed Unbound Plasma Concentration for Mobocertinib and Its Active Metabolites (AP32960 and AP32914)
Time Frame: Day 1 pre-dose and at multiple time points (up to 216 hours) post-dose
Population: PK set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile (e.g., exposure to treatment, availability of measurements and absence of major protocol violations).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Moderate HI (Child-Pugh B): Mobocertinib 40 mg | Severe HI (Child-Pugh C): Mobocertinib 40 mg | Normal Hepatic Function: Mobocertinib 40 mg
Number analyzed (Participants) | 8 | 8 | 8
ng/mL
  Mobocertinib | 0.153 (51.2) | 0.167 (50.3) | 0.184 (39.7)
  AP32960 | 0.0569 (24.4) | 0.0396 (35.9) | 0.0729 (22.2)
  AP32914 | 0.00518 (81.3) | 0.00837 (28.9) | 0.0127 (36.1)

3. Primary Outcome: AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Mobocertinib and Its Active Metabolites (AP32960 and AP32914)
Time Frame: Day 1 pre-dose and at multiple time points (up to 216 hours) post-dose
Population: PK set included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile (e.g., exposure to treatment, availability of measurements and absence of major protocol violations). Number analyzed is the number of participants with data available for analysis for the specified category. Data was not collected for AP32914 as no participant displayed a sufficient PK profile with respect to this parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hours/milliliters (ng*h/mL)
Arm/Group | Moderate HI (Child-Pugh B): Mobocertinib 40 mg | Severe HI (Child-Pugh C): Mobocertinib 40 mg | Normal Hepatic Function: Mobocertinib 40 mg
Number analyzed (Participants) | 8 | 8 | 8
nanogram*hours/milliliters (ng*h/mL)
  Mobocertinib | 206 (32.7) | 291 (48.9) | 199 (36.2)
  AP32960: number analyzed (Participants) | 5 | 2 | 8
  AP32960 | 91.6 (22.2) | 115 (1.94) | 105 (31.5)
  AP32914: number analyzed (Participants) | 0 | 0 | 0

4. Primary Outcome: AUC∞,u: Area Under the Unbound Plasma Concentration-time Curve From Time 0 to Infinity for Mobocertinib and Its Active Metabolites (AP32960 and AP32914)
Time Frame: Day 1 pre-dose and at multiple time points (up to 216 hours) post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Moderate HI (Child-Pugh B): Mobocertinib 40 mg | Severe HI (Child-Pugh C): Mobocertinib 40 mg | Normal Hepatic Function: Mobocertinib 40 mg
Number analyzed (Participants) | 8 | 8 | 8
ng*h/mL
  Mobocertinib | 3.26 (42.6) | 4.31 (42.4) | 3.50 (34.9)
  AP32960: number analyzed (Participants) | 5 | 2 | 8
  AP32960 | 1.32 (28.4) | 1.48 (28.5) | 1.60 (29.3)
  AP32914: number analyzed (Participants) | 0 | 0 | 0

5. Primary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Mobocertinib and Its Active Metabolites (AP32960 and AP32914)
Time Frame: Day 1 pre-dose and at multiple time points (up to 216 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Moderate HI (Child-Pugh B): Mobocertinib 40 mg | Severe HI (Child-Pugh C): Mobocertinib 40 mg | Normal Hepatic Function: Mobocertinib 40 mg
Number analyzed (Participants) | 8 | 8 | 8
ng*h/mL
  Mobocertinib | 192 (34.2) | 275 (50.3) | 186 (38.7)
  AP32960 | 69.3 (21.3) | 64.5 (52.1) | 91.9 (35.1)
  AP32914 | 7.61 (48.1) | 9.32 (91.4) | 12.5 (71.3)

6. Primary Outcome: AUClast,u: Area Under the Unbound Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Mobocertinib and Its Active Metabolites (AP32960 and AP32914)
Time Frame: Day 1 pre-dose and at multiple time points (up to 216 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Moderate HI (Child-Pugh B): Mobocertinib 40 mg | Severe HI (Child-Pugh C): Mobocertinib 40 mg | Normal Hepatic Function: Mobocertinib 40 mg
Number analyzed (Participants) | 8 | 8 | 8
ng*h/mL
  Mobocertinib | 3.04 (43.3) | 4.06 (42.9) | 3.28 (36.2)
  AP32960 | 1.02 (24.9) | 0.906 (42.8) | 1.40 (32.0)
  AP32914 | 0.0524 (82.5) | 0.108 (45.5) | 0.138 (79.5)

7. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Mobocertinib and Its Active Metabolites (AP32960 and AP32914)
Time Frame: Day 1 pre-dose and at multiple time points (up to 216 hours) post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Moderate HI (Child-Pugh B): Mobocertinib 40 mg | Severe HI (Child-Pugh C): Mobocertinib 40 mg | Normal Hepatic Function: Mobocertinib 40 mg
Number analyzed (Participants) | 8 | 8 | 8
hours (h)
  Mobocertinib | 2.00 [1.00 to 8.00] | 4.00 [1.00 to 8.00] | 6.00 [1.00 to 8.00]
  AP32960 | 2.00 [2.00 to 4.00] | 4.00 [2.00 to 6.00] | 6.00 [2.00 to 6.00]
  AP32914 | 5.00 [2.00 to 8.00] | 4.00 [2.00 to 8.00] | 6.00 [2.00 to 8.00]

8. Primary Outcome: t1/2z: Terminal Disposition Phase Half-life for Mobocertinib and Its Active Metabolites (AP32960 and AP32914)
Time Frame: Day 1 pre-dose and at multiple time points (up to 216 hours) post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Moderate HI (Child-Pugh B): Mobocertinib 40 mg | Severe HI (Child-Pugh C): Mobocertinib 40 mg | Normal Hepatic Function: Mobocertinib 40 mg
Number analyzed (Participants) | 8 | 8 | 8
hours
  Mobocertinib | 26.4 (16.8) | 30.7 (20.9) | 22.9 (28.1)
  AP32960: number analyzed (Participants) | 5 | 2 | 8
  AP32960 | 31.7 (36.2) | 45.0 (44.9) | 25.9 (29.1)
  AP32914: number analyzed (Participants) | 0 | 0 | 0

9. Primary Outcome: λz: Terminal Elimination Rate Constant for Mobocertinib and Its Active Metabolites (AP32960 and AP32914)
Description: Terminal elimination rate constant (λz) is a mathematical estimate calculated using log-linear regression of the terminal portions of a plasma concentration against time curve.
Time Frame: Day 1 pre-dose and at multiple time points (up to 216 hours) post-dose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Moderate HI (Child-Pugh B): Mobocertinib 40 mg | Severe HI (Child-Pugh C): Mobocertinib 40 mg | Normal Hepatic Function: Mobocertinib 40 mg
Number analyzed (Participants) | 8 | 8 | 8
1/hour
  Mobocertinib | 0.0263 (16.8) | 0.0226 (20.9) | 0.0303 (28.1)
  AP32960: number analyzed (Participants) | 5 | 2 | 8
  AP32960 | 0.0218 (36.2) | 0.0154 (44.9) | 0.0268 (29.1)
  AP32914: number analyzed (Participants) | 0 | 0 | 0

10. Primary Outcome: CL/F: Apparent Clearance After Extravascular Administration for Mobocertinib
Time Frame: Day 1 pre-dose and at multiple time points (up to 216 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour (L/hour)
Arm/Group | Moderate HI (Child-Pugh B): Mobocertinib 40 mg | Severe HI (Child-Pugh C): Mobocertinib 40 mg | Normal Hepatic Function: Mobocertinib 40 mg
Number analyzed (Participants) | 8 | 8 | 8
liters per hour (L/hour) | 195 (32.7) | 137 (48.9) | 201 (36.2)

11. Primary Outcome: CLu/F: Apparent Clearance for Unbound Drug After Extravascular Administration for Mobocertinib
Time Frame: Day 1 pre-dose and at multiple time points (up to 216 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hour
Arm/Group | Moderate HI (Child-Pugh B): Mobocertinib 40 mg | Severe HI (Child-Pugh C): Mobocertinib 40 mg | Normal Hepatic Function: Mobocertinib 40 mg
Number analyzed (Participants) | 8 | 8 | 8
L/hour | 12300 (42.6) | 9290 (42.4) | 11400 (34.9)

12. Primary Outcome: Vz/F: Apparent Volume of Distribution During the Terminal Disposition Phase After Extravascular Administration for Mobocertinib
Time Frame: Day 1 pre-dose and at multiple time points (up to 216 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Moderate HI (Child-Pugh B): Mobocertinib 40 mg | Severe HI (Child-Pugh C): Mobocertinib 40 mg | Normal Hepatic Function: Mobocertinib 40 mg
Number analyzed (Participants) | 8 | 8 | 8
liters | 7400 (30.5) | 6090 (30.7) | 6640 (37.7)

13. Primary Outcome: Vz,u/F: Apparent Volume of Distribution for Unbound Drug During the Terminal Disposition Phase After Extravascular Administration for Mobocertinib
Time Frame: Day 1 pre-dose and at multiple time points (up to 216 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Moderate HI (Child-Pugh B): Mobocertinib 40 mg | Severe HI (Child-Pugh C): Mobocertinib 40 mg | Normal Hepatic Function: Mobocertinib 40 mg
Number analyzed (Participants) | 8 | 8 | 8
liters | 467000 (34.3) | 412000 (22.6) | 377000 (24.9)

14. Secondary Outcome: Plasma Protein Binding of Mobocertinib and Its Active Metabolites (AP32960 and AP32914)
Time Frame: Day 1 at multiple time points (up to 24 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage bound
Arm/Group | Moderate HI (Child-Pugh B): Mobocertinib 40 mg | Severe HI (Child-Pugh C): Mobocertinib 40 mg | Normal Hepatic Function: Mobocertinib 40 mg
Number analyzed (Participants) | 8 | 8 | 8
percentage bound
  Mobocertinib | 98.4 (0.385) | 98.5 (0.397) | 98.2 (0.426)
  AP32960 | 98.5 (0.114) | 98.6 (0.321) | 98.5 (0.129)
  AP32914 | 99.2 (0.332) | 98.7 (0.621) | 98.9 (0.245)

15. Secondary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant administered a pharmaceutical product; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (e.g., a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Baseline up to 30 days after last dose of study drug (up to Day 32)
Population: Safety set included all participants who received the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate HI (Child-Pugh B): Mobocertinib 40 mg | Severe HI (Child-Pugh C): Mobocertinib 40 mg | Normal Hepatic Function: Mobocertinib 40 mg
Number analyzed (Participants) | 8 | 8 | 8
Participants | 1 | 0 | 2

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after last dose of study drug (up to Day 32)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Safety set included all participants who received the study drug.
Arm/Group | Moderate HI (Child-Pugh B): Mobocertinib 40 mg | Severe HI (Child-Pugh C): Mobocertinib 40 mg | Normal Hepatic Function: Mobocertinib 40 mg
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 0/8 | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Moderate HI (Child-Pugh B): Mobocertinib 40 mg (N=8) | Severe HI (Child-Pugh C): Mobocertinib 40 mg (N=8) | Normal Hepatic Function: Mobocertinib 40 mg (N=8)
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2020-08-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT04056468/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT04056468/SAP_001.pdf